CLINICAL TRIAL: NCT06242015
Title: The Effect of Ordered Eating on Postprandial Glucose and Substrate Utilization During an Acute Exercise Bout
Brief Title: Ordered Eating and Acute Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Patrick Wilson, PhD, Associate Professor of Exercise Science, Old Dominion University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 24-003
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Glucose Metabolism Disorders; Hunger
Keywords: Exercise; Glucose; Fat metabolism; Hunger
MeSH Terms: conditions — Glucose Metabolism Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbohydrate-first meal (Experimental)
  Interventions: Other: Carbohydrate-first meal
- Carbohydrate-last meal (Experimental)
  Interventions: Other: Carbohydrate-last meal

INTERVENTIONS:
Other: Carbohydrate-first meal — Rice (150 grams) eaten first, followed by broccoli (150 grams) and chicken (100 grams)
  Arms: Carbohydrate-first meal
Other: Carbohydrate-last meal — Broccoli (150 grams) and chicken (100 grams) eaten first, followed by rice (150 grams)
  Arms: Carbohydrate-last meal

SUMMARY:
There is well documented evidence that ingesting dietary carbohydrate in large amounts tends to increase postprandial glucose. In healthy populations, this is not necessarily a problem, but continuous exposure to high levels of glucose-hyperglycemia-is a defining characteristic and risk factor for type 2 diabetes mellitus. Consuming a carbohydrate-rich food as the final food in a meal sequence has been shown to significantly reduce postprandial glucose excursions in both diabetes patients and in healthy controls. The exact mechanisms behind this phenomenon are not well understood, but one proposed course is simply that the vegetable and protein already being digested slows the rate of glucose rise.

Despite the findings, little-to-no research has examined how manipulating the order of foods in a meal impacts subsequent exercise responses. In this experimental crossover study, each participant will undergo two acute feeding conditions (carbohydrate-rich foods first vs. last in a meal), which will be followed by exercise 60 minutes later. We will observe the effects of meal order on postprandial glucose, substrate/fuel utilization, and subjective perceptions at rest and during 30 minutes of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Currently physically active (scheduled exercise at least three days per week for 30 minutes each time over the last three months)
* Ability to perform moderate-to-high intensity running for at least 30 minutes

Exclusion Criteria:

* Any allergy or other condition that would prohibit the consumption of poultry, rice, or broccoli
* Any injury or disease (cardiovascular disease, diabetes, pulmonary disease except controlled asthma) precluding physical exercise
* Currently pregnant
* Implanted electrical devices such as a pacemaker.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose | 2 hours (premeal and 30, 60, 90, and 120 minutes after eating)
  Blood glucose will be measured with fingerstick samples and a portable glucometer

SECONDARY OUTCOMES:
Carbohydrate use | 100 minutes (premeal and continuously for 90 minutes after eating)
  Carbohydrate utilization will be estimated from respiratory gas exchange
Fat use | 100 minutes (premeal and continuously for 90 minutes after eating)
  fat utilization will be estimated from respiratory gas exchange
Hunger-satiety perceptions | 2 hours (Premeal and at 15, 30, 45, 60, 68, 78, 88, 120 minutes after eating)
  Hunger, appetite, satiety, and fullness on a 0-10 Likert scale
Rating of perceived exertion | 30 minutes (at 8, 18, 28 minutes of exercise)
  Rating of effort during 30-minute exercise bout

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wilson, Principal Investigator — Old Dominion University
Locations (1):
- ODU Human Performance Laboratory, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared upon reasonable request. Requests should be made to the corresponding author.
Time Frame: The data will be made available upon the study's publication and will remain available for at least 5 years
Access Criteria: Researchers with a justified reason for wanting access to the data